CLINICAL TRIAL: NCT00379366
Title: Efficacy and Tolerance of Transcutaneous Ionizing Radiations to Prevent Restenosis Caused by Intimal Hyperplasia on Prosthetic Haemodialysis Vascular Access
Brief Title: External Ionizing Radiation to Prevent Restenosis on Haemodialysis Vascular Access
Acronym: RASTA
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: lack of patients
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9443-05; 2005-011
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Renal Insufficiency, Chronic; Graft Occlusion, Vascular; Thrombosis; Intimal Hyperplasia
Keywords: Randomized Controlled Trials; Renal Dialysis; Graft Occlusion, Vascular; Angioplasty; Vascular Patency; Radiation, Ionizing
MeSH Terms: conditions — Renal Insufficiency, Chronic; Graft Occlusion, Vascular; Thrombosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 14 Gy ionizing radiations
  Interventions: Device: External ionizing radiations
- 2 (No Intervention)

INTERVENTIONS:
Device: External ionizing radiations — 14 Gy in one time
  Arms: 1

SUMMARY:
Although ionizing radiations have been proposed for the prevention of intimal hyperplasia in coronary and peripheral arteries, information is lacking on how irradiation may prevent neointimal smooth-muscle cell proliferation and restenosis on prosthetic haemodialysis vascular access. We will assess the preventive effect of one dose of radiations (14 Gy) administered transcutaneously one day after dilatation of stenosis on prosthetic haemodialysis vascular access in a randomized controlled trial with a standardized clinical and ultrasonographic one-year follow-up.

DETAILED DESCRIPTION:
Background: one of the major clinical concerns of prosthetic haemodialysis access is the risk of possible restenosis after stenosis dilatation. Only 25% of dilated prosthetic haemodialysis vascular accesses remain patent at one year. No available pharmacological agents can yet effectively prevent it. After stenosis dilatation the vascular wall responds to mechanical injury in a standardized manner: intimal smooth-muscle cells migrate and proliferate, a neointima gradually begins to form and the cell phenotype changes from contractile to secretory. One way to inhibit the neointimal proliferation responsible for restenosis is to induce cell apoptosis by delivering ionizing radiations to the dilated area after the endovascular procedure. Experimental studies and multicenter clinical trials have reported the beneficial effects of endovascular beta or gamma ionizing radiation on vascular restenosis. Experimental studies in animals and recent clinical trials clearly show that external irradiation also reduces neointimal proliferation after arterial injury thus opening the way for the clinical assessment of ionizing radiations on arteries. In a previous experimental study, we reported that irradiation has a dose-dependent effect on the prevention of restenosis: a dose larger than 10 Gy is needed to obtain a significant reduction of intimal hyperplasia.

Objective: the main objective is to assess external ionizing radiation for restenosis prevention on prosthetic haemodialysis vascular accesses after angioplasty. A secondary objective is to assess the treatment safety.

Methods: Single blind randomized clinical trial on two parallel groups of 53 patients each. Patients with chronic renal failure treated by dialysis will be included after a successful angioplasty on a stenosis of the vein adjacent to their prosthetic haemodialysis vascular access. One group will be treated by a single dose of ionizing radiations (14 Gy) at day 1 after angioplasty. The control group will not receive any preventive treatment. The primary outcome is the one-year vascular access patency failure. Secondary outcomes are the one-year delay of occurrence of a restenosis and the treatment safety. Outcomes will be assessed by a clinical and ultrasonographic (at 1, 3, 6 and 12 months, or at other time points in case of stenosis suspicion) follow-up.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years
* successful angioplasty (residual stenosis < 30%) on a significant stenosis (maximal systolic speed 3 times > from basal maximal systolic speed, stenosis > 70% on angiography) on the venous-prosthesis anastomosis or on the venous segment 5 cm after the anastomosis of a prosthetic haemodialysis vascular access (at least 1 month old)
* social security affiliation
* signed informed consent

Exclusion Criteria:

* contra-indications of radiotherapy
* angioplasty with stenting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Thrombosis or stenosis > to 70% or indication of a new treatment of stenosis during the 12 month follow-up | 1, 3, 6 and 12 month after initial angioplasty

SECONDARY OUTCOMES:
Stenosis (> to 70%) or thrombosis or indication of a new treatment occurring | 1, 3, 6 or 12 months after initial angioplasty
safety | 1, 3, 6 and months after initial angioplasty

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe MAIRE, Pr, Principal Investigator — University Hospital, Bordeaux, France; Paul Perez, Dr, Study Chair — University Hospital, Bordeaux, France
Locations (5):
- France (5):
  - Clinc Delay, Bayonne
  - Côte Basque Hospital, Bayonne
  - Clinic Saint Augustin, Bordeaux
  - Service de Chirurgie Vasculaire, Hôpital Pellegrin-tripode, CHU de Bordeaux, Bordeaux
  - Clinic Francheville, Périgueux